CLINICAL TRIAL: NCT05733065
Title: A Study of the Placental Methylome of Dichorionic and Monochorionic Monozygotic Twin Pairs to Establish a Timeline of Epigenetic Programming
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC-08264
Record Dates: First submitted 2021-01-26; First posted 2023-02-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Twin Placenta
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monozygotic Twin (Other): we will include natural conceived twin pairs born before 2002, with known birth weight, sex and gestational age, and where both twins were live born without congenital abnormality. Twins born after pregnancies complicated by conditions such as TTTS will be excluded. MZ twins pairs will be ranked according to intra-pair birth weight difference. Next, we intend to include the 120 most discordant monozygotic twin pairs, stratified by chorionicity (1:1 ratio) and in the case of DC by fusion of the placentas (1:1 ratio). Only pairs where both twins consent to inclusion in the study will be included.
  Interventions: Other: saliva sample; Other: questionnaire

INTERVENTIONS:
Other: saliva sample — Adult twins will be asked to send saliva samples in a reply envelope to Maastricht University, department of Genetics and Cell Biology, where they will be frozen and stored before analysis. DNA will be extracted from the saliva using a commercially available kit according to the manufacturer's instructions.
Other: questionnaire — Along with saliva samples, adult twins, will be asked to complete a questionnaire about their health. Study subjects will be asked to self-report height and weight. Additionally, questions will focus on cardiometabolic risk, including questions about smoking, physical activities, medical diagnoses, current medications, family history of cardiometabolic disease, and for female twins an obstetric and gynaecological history, including number of pregnancies and pregnancy complications (such as gestational diabetes and pre-eclampsia). The questionnaire will take the form of a self-completed, web-based questionnaire which will be hosted by the Qualtrics platform (Qualtrics.com). This platform is supported by the University of Maastricht due to its security and privacy measures.

SUMMARY:
The timing of the moment of splitting is variable amongst twins and can be inferred from chorionicity, allowing a time-line of early environmental influences to be established. Monozygotic twins can remain discordant for growth and health outcomes throughout life, implying the prenatal establishment of a regulatory program with effects that persist into adulthood.

Objective: To investigate the effect of the moment of splitting (chorionicity) on the placental and saliva (in adulthood) methylome and cardiometabolic disease risk in monozygotic twin pairs. Birth weight discordance will be used as an indicator of prenatal environmental heterogeneity between the twins.

DETAILED DESCRIPTION:
Rationale: The developmental origins of health and disease (DoHaD) hypothesis, states that antenatal and early life exposure to a suboptimal environment can predispose for adverse health outcomes in adult life, such as cardiometabolic disease. Modification of the epigenome, and more specifically the methylome, seems a plausible mechanism for this. It has been shown that a suboptimal early environment, such as famine during the periconception period, can perturb DNA methylation signatures of the offspring. Furthermore, the preimplantation period is likely to represent a critical window for the establishment of optimal DNA methylation as epigenetic reprogramming takes place during this time. The precise influence of environmental factors during this time is incompletely understood; human studies of the preimplantation period are complicated by an inaccessibility of samples and the high variability of the environment induced by maternal factors. Here, the study of monozygotic twins can be employed. Although monozygotic twins are genetically identical, they can differ phenotypically, for example in birth weight. Phenotype and methylome differences attributable to genetic and maternal differences can be ruled out, meaning that intra-pair differences must be a result of variation in their prentatal environment. Furthermore, the moment of splitting defines the point from which twins can experience environmental differences. The timing of the moment of splitting is variable amongst twins and can be inferred from chorionicity, allowing a time-line of early environmental influences to be established. Monozygotic twins can remain discordant for growth and health outcomes throughout life, implying the prenatal establishment of a regulatory program with effects that persist into adulthood.

Objective: To investigate the effect of the moment of splitting (chorionicity) on the placental and saliva (in adulthood) methylome and cardiometabolic disease risk in monozygotic twin pairs. Birth weight discordance will be used as an indicator of prenatal environmental heterogeneity between the twins.

Study design: prospective twin cohort - using a subset of twins from the East Flanders Prospective Twin Study (EFPTS).

Main study parameters/endpoints: Placenta (birth) and saliva (adulthood) DNA methylation. Questionnaire-based adult anthropometric measurements and cardiometabolic disease risk data.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no risk or benefit to participants associated with participation in this study as DNA methylation analyses cannot be used to identify disease (susceptibility). Placental tissue samples were already collected at birth and stored in a biobank. Further samples for DNA methylation analysis will be collected non-invasively by saliva sample. There is a minor time burden associated with participation in questionnaire-based data collection at the adult time point, however this is not expected to be excessive.

ELIGIBILITY:
Inclusion Criteria:

* natural conceived twin pairs born before 2002,
* with known birth weight, sex and gestational age,
* where both twins were live born without congenital abnormality
* Only pairs where both twins consent to inclusion in the study will be included.

Exclusion Criteria:

* Twins born after pregnancies complicated by conditions such as TTTS will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify differences in DNA methylation in placental biopsy. | 1 year after saliva sample collection
  Placental DNA extraction will be carried out using a commercially available kit such as QIAamp DNA Mini Kit. We will first identify differences in placental DNA methylation that are associated with time-of splitting, i.e. chorionicity, to identify epigenome alterations that are attributable to the preimplantation period. Thereafter, birth weight discordance (weight of the heaver twin minus weight of the lighter twin, divided by weight of the heavier twin, multiplied by 100) will be used as a measure of antenatal environmental differences between the twins to identify loci of differential methylation that relate to environmental differences experienced in early gestation.
To identify differences in DNA methylation in saliva sample. | 1 year after saliva sample collection
  Adult twins will be asked to send saliva samples. DNA will be extracted from the saliva using a commercially available kit. The adult methylome, deduced from saliva, will be interrogated to determine whether the methylation signatures associated with differences in the early embryonic environment persist into adulthood.

SECONDARY OUTCOMES:
To identify epigenetic alterations, present at birth that persist into adulthood, and predict growth/cardiometabolic disease risk parameters. | 1 year after saliva sample collection
  The adult outcomes, such as anthropometric measures and cardiometabolic disease risk factors, obtained from questionnaires will be used to develop a prediction model. The model will take into account biological data collected at birth as well as the placental methylome to predict growth and cardiometabolic outcomes in adulthood. For this purpose we will use techniques such as random forests, which use a fully annotated training dataset to classify subjects. Subsequently, further data points can be entered into the model, and will be assigned to the class that they most closely resemble.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University hospital, Ghent, Belgium